CLINICAL TRIAL: NCT02708121
Title: Increasing Uptake of Behavioral Weight Loss Programs Among Primary Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB201701301-N; 1K23HL127334 (NIH); Pro00079803 (Other: Duke Unversity)
Record Dates: First submitted 2016-03-10; First posted 2016-03-15 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Staff recruiting participants and doing outcomes assessment will remain blinded to treatment assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Participant receives intervention to motivate weight loss treatment initiation and access to weight loss treatment.
  Interventions: Behavioral: Motivational Intervention
- Comparator Arm (Active Comparator): Participant receives access to weight loss treatment alone.
  Interventions: Other: Comparator Intervention

INTERVENTIONS:
Behavioral: Motivational Intervention — Participants complete web-based assessment and receive tailored feedback to motivate weight loss treatment initiation and informed that they have access to weight loss treatment.
  Other Names: Your Wellness Prescription
  Arms: Intervention arm
Other: Comparator Intervention — Participants informed that they have access to weight loss treatment.
  Arms: Comparator Arm

SUMMARY:
This pilot trial will test feasibility and acceptability of a primary care-based intervention that aims to increase the portion of patients who enter evidence-based behavioral weight loss treatment.

DETAILED DESCRIPTION:
This trial is a pilot, pragmatic cluster randomized trial conducted in primary care clinics to determine intervention acceptability and the feasibility of proposed study protocol.

ELIGIBILITY:
Primary care provider Inclusion criteria:

* Employed by Duke PCRC clinic as primary care provider at least ½ FTE.
* Has a primary adult panel
* Has worked at Duke PCRC clinic for at least one year

Patient inclusion criteria

* BMI ≥ 30 kg/m2 as measured at any clinic in previous 12 months.
* English speaking
* Self-report BMI ≥ 29 kg/m2 (to allow for under-reporting)
* Regular email usage, defined as accessing email 3 or more times per week (on home or work computer or cell phone)
* Age 18-75
* Clinical appointment (well visit or chronic care visit) with enrolled Duke provider in 2-6 weeks of record review.
* At least one prior appointment with the provider they are scheduled to see at target clinical appt.
* Has a valid email address in electronic health records.

Patient exclusion criteria:

* In weight loss treatment program in past year
* Unable to read content on websites without any assistance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-03-03 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan A McVay, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] McVay MA, Yancy WS, Bennett GG, Levine E, Jung SH, Jung S, Anton S, Voils CI. A web-based intervention to increase weight loss treatment initiation: results of a cluster randomized feasibility and acceptability trial. Transl Behav Med. 2021 Feb 11;11(1):226-235. doi: 10.1093/tbm/ibz143. PMID 31586443

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All six providers who were recruited through a Duke Health primary care-based research network and were present at a primary care clinic provider meeting in February 2017, were eligible and consented to participate. Patients of the enrolled providers were recruited from May 2017 to August 2017 through an electronic health record database search.
Pre-assignment Details: None of the providers were withdrawn from the study. Of the 66 patients initially consented, 6 withdrew prior to learning their randomization assignment; 4 chose to withdraw for no stated reason; one was withdrawn by the study team due to being in treatment; and one was withdrawn by the study team due to canceling their index appointment.
Groups:
- Mobilization Tool Arm: Participant receives intervention to motivate weight loss treatment initiation and access to weight loss treatment.
  Motivational Intervention: Participants complete web-based assessment and receive tailored feedback to motivate weight loss treatment initiation and informed that they have access to weight loss treatment.
- Comparator Tool Arm: Participant receives access to weight loss treatment alone.
  Comparator Intervention: Participants informed that they have access to weight loss treatment.
Period: Overall Study
Arm/Group | Mobilization Tool Arm | Comparator Tool Arm
Started | 35 | 31
Provided Acceptability Data (No. of participants who completed the post mobilization tool acceptability survey.) | 20 | 0 (This condition did not participate in acceptability survey)
Treatment Program Use Data Available (No. of participants in which the treatment program provided initiation data) | 34 | 24
6 Month In-Person Follow Up Data (No. of participants who attended the six month assessment follow up) | 22 | 19
6 Month Weight Data Via EHR (No. of participants in which their weight data at 6 month follow up was available via health record) | 14 | 13
Completed (No. of participants who received allocated intervention) | 34 | 26
Not Completed | 1 | 5
Not completed — Withdrawn by Study Team | 1 | 1
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Population: One patient in the Comparator Arm completed the screener questionnaire but did not attend baseline session. Thus data is presented for 25 of the 26 enrolled patients for all variable except gender.
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobilization Tool Arm | Comparator Tool Arm | Total
Number analyzed (Participants) | 34 | 26 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One patient in the Comparator Arm completed the screener questionnaire but did not attend baseline session. Thus data is presented for 25 of the 26 enrolled patients for all variable except gender.
  years
    number analyzed (Participants) | 34 | 25 | 59
    (all) | 54.4 (14.0) | 54.9 (10.9) | 54.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 34
  Male | 15 | 11 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: One patient in the Comparator Arm completed the screener questionnaire but did not attend baseline session. Thus data is presented for 25 of the 26 enrolled patients for all variable except gender.
  Participants
    White, Non-Hispanic: number analyzed (Participants) | 34 | 25 | 59
    White, Non-Hispanic | 23 | 16 | 39
    African American: number analyzed (Participants) | 34 | 25 | 59
    African American | 10 | 9 | 19
    Other or multiple races: number analyzed (Participants) | 34 | 25 | 59
    Other or multiple races | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Attending 6 Month Follow-up Appointment
Description: Count of enrolled participants who attend 6 month follow-up appointment
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mobilization Tool Arm | Comparator Tool Arm
Number analyzed (Participants) | 34 | 26
Participants | 22 | 19

2. Secondary Outcome: Intervention Acceptability (Acceptability Outcome)
Description: Ratings on series of items developed by study team to assess patient perception of acceptability of the intervention. Items were created by study team. Possible range of 1 (strongly disagree) to 5 (strongly agree). Higher score reflects greater acceptability except for item 11.
Time Frame: 1 month
Population: Among mobilization tool participants, 28 patients progressed past the tool's introductory page, and 27 patients completed the tool. The post-tool acceptability survey was completed by 20 participants (72% of those who began the tool).
Measure: Mean (Standard Deviation); unit: score on a item
Arm/Group | Mobilization Tool Arm
Number analyzed (Participants) | 20
score on a item
  Item 1: Enjoyed | 4.15 (0.67)
  Item 2: Learning | 4.05 (0.83)
  Item 3: Easy to use | 4.25 (0.72)
  Item 4: Secure | 4.30 (0.73)
  Item 5: Interested | 4.10 (0.72)
  Item 6: Trustworthy | 4.15 (0.75)
  Item 7: Enough time | 4.15 (0.75)
  Item 8: Easy to understand | 4.35 (0.59)
  Item 9: Easy to navigate | 4.40 (0.50)
  Item 10: Useful | 4.15 (0.67)
  Item 11: Too long | 2.45 (1.39)
  Item 12: Enough information | 4.10 (0.64)

3. Other Pre Specified Outcome: Number of Participants Who Initiated Treatment Based on Program-provided Data and Self-report
Description: Number of participants who initiate evidence-based weight loss treatment. Initiation is defined as completing at least one session (either group in-person session, one-on-one)
Time Frame: 6 months
Population: Six participants withdrew prior to learning randomization condition and were not followed.
Measure: Count of Participants; unit: Participants
Arm/Group | Mobilization Tool Arm | Comparator Tool Arm
Number analyzed (Participants) | 34 | 26
Participants
  Treatment initiation, program data: number analyzed (Participants) | 34 | 24
  Treatment initiation, program data | 20 | 8
  Treatment initiation, self-report: number analyzed (Participants) | 22 | 19
  Treatment initiation, self-report | 14 | 8

ADVERSE EVENTS:
Time Frame: 6 months (study period)
Arm/Group | Mobilization Tool Arm | Comparator Tool Arm
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/34 | 0/26
Other Adverse Events (participants affected / at risk) | 0/34 | 0/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mobilization Tool Arm (N=34) | Comparator Tool Arm (N=26)
Hospitalization (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant was not hospitalized due to intervention.

LIMITATIONS AND CAVEATS:
A fully powered trial is needed to test intervention effectiveness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT02708121/Prot_SAP_000.pdf